CLINICAL TRIAL: NCT06903468
Title: Novel Cavity Marking Technique in Breast Cancer Patients Undergoing Breast Conservation Surgery With Oncoplastic Reconstruction for the Delivery of Adjuvant Radiotherapy and Accuracy of Recommended Re-excisions
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UF-BRE-015; IRB202500675 (Other: University of Florida)
Record Dates: First submitted 2025-03-24; First posted 2025-03-30 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Ductal Carcinoma in Situ; Breast Cancer
Keywords: invasive breast cancer; non-invasive ductal carcinoma in-situ; oncoplastic reconstruction; breast conservation surgery; boost volume; cavity marking; breast
MeSH Terms: conditions — Carcinoma, Intraductal, Noninfiltrating; Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Novel cavity marking technique during breast conservation surgery with oncoplastic reconstruction (Experimental)
  Interventions: Procedure: Novel cavity marking technique

INTERVENTIONS:
Procedure: Novel cavity marking technique — A novel cavity marking technique will be performed on all participants during their breast conservation surgery. For this technique, cavity marking will be in a clockwise fashion per breast starting with the superior margin of the tumor bed. The superior margin of the left breast will be marked with a single large clip, followed by a double clip for the lateral margin, a triple clip for the inferior margin, and a quadruple clip for the medial margin. The superior margin of the right breast will be marked with a single large clip, followed by a double clip for the medial margin, a triple clip for the inferior margin and a quadruple clip for the lateral margin. Margins with multiple clips will always have one large clip with the remaining clips standard medium size.

SUMMARY:
This study will investigate a novel approach to marking surgical cavity margins following tumor resection, to allow for more accurate radiotherapy following oncoplastic surgery. Our proposed cavity marking schema will allow radiation oncology to identify the cavity margins more accurately on CT simulation for radiation planning and delivery. This cavity marking schema also provides more accurate margin identification in patients recommended for re-excision of close or positive margins.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 18 years of age.
* A pathological diagnosis consistent with non-invasive ductal carcinoma in-situ (DCIS) and invasive breast cancer, Tis-T3N0-3M0
* Subject is planning to undergo or has undergone breast conservation surgery and oncoplastic reconstruction with cavity marking surgery.
* ECOG Performance status of 0-1
* Written informed consent obtained from the subject and the subject agrees to comply with all the study-related procedures.
* Subjects must not have more than one active malignancy at the time of enrollment (Subjects with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen [as determined by the treating physician or approved by the PI] may be included).
* Subjects of childbearing potential (SOCBP) must be using an adequate method of contraception to avoid pregnancy during surgery and radiation therapy. Prior to study enrollment, subjects of childbearing potential must be advised of the importance of avoiding pregnancy during the surgery and radiation portions of the trial and the potential risk factors for an unintentional pregnancy. SOCBP includes any subject who has experienced menarche and who has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or who is not post-menopausal. Post-menopause is defined as amenorrhea that has lasted for ≥ 12 consecutive months without another cause.

Exclusion Criteria:

* Patient not recommended for, or have declined, adjuvant radiotherapy
* Subjects with prior ipsilateral breast surgery and identifiable surgical clips.
* Subjects who are confirmed to be pregnant or breastfeeding.
* History of any other disease, metabolic dysfunction, clinical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of protocol therapy or that might affect the interpretation of the results of the study or that puts the subject at high risk for treatment complications, in the opinion of the treating physician.
* Prisoners or subjects who are involuntarily incarcerated, or subjects who are compulsorily detailed for treatment of either a psychiatric or physical illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-10-27 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2029-11 (Estimated)

PRIMARY OUTCOMES:
Confidence rating in cavity identification | Within 8 weeks of surgery if patient does not receive adjuvant chemotherapy or within 8 weeks following adjuvant chemotherapy (~4-6 months after surgery
  Determine the percentage of patients that receive each of three possible confidence ratings ("Confident", "Informative", and "Ambiguous") from radiation oncologists for their confidence in being able to identify the surgical cavity on imaging.

SECONDARY OUTCOMES:
Percent of patients needing re-excision | 7-14 days post-surgery
  Determine the percentage of patients needing re-excision
Local disease recurrence rate | 2 years post-surgery
  Determine the percentage of patients that have local disease recurrence at 2 years post-surgery
Median overall survival rate | 2 years post-surgery
  Determine the median overall survival rate at 2 years post-surgery.
Median recurrence-free survival rate | 2 years post-surgery
  Determine the median recurrence-free survival rate at 2 years post-surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Spiguel, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States